CLINICAL TRIAL: NCT05234034
Title: Intensity of Physical Activity Level During Daily Living: Unravelling Its Relationship With Chronic Musculoskeletal Disorders and Evaluating Underlying Facilitators and Barriers, An Exploratory Survey Study
Acronym: MSK-SUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Associate Professor, Hasselt University
Other Study IDs: B1152021000021
Record Dates: First submitted 2022-01-17; First posted 2022-02-10 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Chronic Musculoskeletal Disease; Exercise Intensity; Physical Activity; Online Survey
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- chronic low back pain (LBP): persons with chronic low back pain (LBP) will be included in this arm.
  Interventions: Other: online survey
- chronic neck pain (CNP): persons with chronic neck pain (CNP) will be included in this arm.
  Interventions: Other: online survey
- chronic shoulder pain (CSP): persons with chronic shoulder pain (CSP) will be included in this arm.
  Interventions: Other: online survey
- osteoarthritis (OA): persons with osteoarthritis (OA) will be included in this arm.
  Interventions: Other: online survey
- fibromyalgia (FM): persons with fibromyalgia (FM) will be included in this arm.
  Interventions: Other: online survey
- chronic Temporomandibular Disorder (CTMD): persons with chronic temporomandibular disorder (CTMD) will be included in this arm.
  Interventions: Other: online survey

INTERVENTIONS:
Other: online survey — participantion consists of filling in an online survey that will take approximately 53 minutes. An adapted battery of questionnaires is provided for each subgroup.

SUMMARY:
chronic musculoskeletal disorders (CMDs) are a hugh burden to healthcare wordwide. Physical activity can improve outcomes related with CMDs, however dose response relationships are poorly understood. Therefore, to date it has not been possible to formulate general recommendations on optimal therapeutic quantity of physical activity. Furthermore, a complexity of possible facilitators and barriers has been stated to limit effective improvement of physical activity in therapy and currently applied low to moderate exercise intensities in rehabilitation could be below the required level to achieve optimal therapy outcomes.

The primary objective of this study is to get insight on the impact of the intensity of the physical activity level on pain and disability in persons with CMDs. Second, the underlying facilitators and barriers to perform physical activity (at different intensities) during daily living will be evaluated. Third, the impact of the intensity of the physical activity level on the motivation to perform a rehabilitation program will be evaluated.

DETAILED DESCRIPTION:
Chronic musculoskeletal disorders (CMDs) affect up to 20% of all persons worldwide, and their prevalence continues to rise steadily. They can have a major impact on the individual as they significantly affect both physical and psychological functioning. As such, they often produce recurring healthcare costs and cause limitations of participation in society and long-term absenteeism. Ultimately, CMDs can be pervasive medical problems and consume huge amounts of healthcare resources.

A key public health intervention recommended for improving health related outcomes of nearly all chronic disorders is physical activity. High level evidence showing beneficial effects of physical activity is also available for multiple CMDs including chronic low back pain, neck pain, and fibromyalgia. Hereby, increased levels of physical activity have been found to improve outcomes such as pain intensity, functional disability, quality of life, mortality risk, and working ability. However, dose-response relationships between physical activity and these therapeutic outcomes are still poorly understood. While an inverse association between low physical activity and increased prevalence of musculoskeletal disorders seems to exist, results of therapeutic programs aimed at increasing physical activity remain contradictory when it comes to improving pain and disability specifically (which might be seen as primary therapy success outcomes for this population). Therefore, to date it has not been possible to formulate general recommendations on optimal therapeutic quantity of physical activity and how activities of daily life should be designed for specific CMD patient populations. Also, although physical activity has clear advantages, it seems difficult to effectively improve physical activity levels of persons with CMDs. A complexity of possible facilitators (e.g. "improved health state", "social support", and "facilitating cognitions, emotions, and behavior") and barriers (e.g. "time restrictions", "social barriers", "maladaptive cognitions, emotions and behavior", and "access to exercise opportunities") has been stated. To accommodate these facilitators and barriers, therapy programs should be sufficiently adapted to the specific needs of the participant.

Exercise therapy is consistently advocated as a primary treatment approach to further support increasing physical activity. However, overall therapy effects also remain low for this training modality. With regard to better adapting this treatment strategy, it has been suggested that the currently applied low to moderate exercise intensities in rehabilitation could be below the required level and that this might attenuate therapy outcomes. Moreover, if persons with CMDs already perform physical activity at a high intensity during their daily living, they might not be motivated to follow low or moderate intensity programs. Besides, setting up a high intensity training (HIT) program can be very valuable to increase therapy success, as HIT programs have already been found to improve outcomes more than comparable programs at moderate intensity in certain MSDs such as chronic low back pain and spondyloarthritis. Nonetheless, on the other hand, persons with other specific types of CMDs, or with a low activity level, might not feel the urge, have the self-confidence, or be deterred to start and persevere in a rehab program with these characteristics.

The primary objective of this study is to get insight on the impact of the intensity of the physical activity level on pain and disability in persons with CMDs. Second, the underlying facilitators and barriers to perform physical activity (at different intensities) during daily living will be evaluated. Third, the impact of the intensity of the physical activity level on the motivation to perform a rehabilitation program will be evaluated.

Primary research question and hypothesis Question 1: to which extent does the intensity level of physical activity during daily living explain variance in outcomes related to pain and functional disability in persons with CMDs?

• Hypothesis 1: Higher pain and higher disability levels are seen in persons with CMDs with lower intensity physical activity levels during daily living.

Secondary research questions and hypotheses Question 2: to which extent are outcomes with regard to psychological factors related to the intensity level of physical activity during daily living in persons with CMDs? • Hypothesis 2: psychological factors have a significant relationship to the activity level of persons with CMDs.

Question 3: Which are the facilitators and barriers for having a moderate or vigorous intensity during daily life physical activity in persons with CMDs?

• Hypothesis 3: Specific facilitators and barriers can be summarized with regard to having a moderate or vigorous intensity physical activity level in persons with CMDs.

Question 4: To which extent does a relationship exist between pain, functional disability, and mediating psychological factors on the one hand and facilitators and barriers for having a moderate or vigorous intensity level of physical during daily living on the other hand in persons with CMDs? • Hypothesis 4: pain, functional disability, and mediating patient characteristics are related to specific facilitators and barriers for a moderate or vigorous intensity level of physical activity during daily living in persons with CMDs.

Question 5: To which extent does the intensity level of physical activity level during daily living relate to motivation to start an exercise therapy program at high intensity?

• Hypothesis 5: Persons with CMDs with a high level of physical activity during daily living will showcase higher motivation to start a therapy program at high intensity.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* A medical diagnosis of one of the following musculoskeletal disorders: chronic low back pain (LBP); chronic neck pain (NP); chronic shoulder pain (CSP); osteoarthritis (OA); chronic Temporomandibular Disorder (CTMD); fibromyalgia (FM).
* Chronic pain, defined as: pain that persists or recurs for longer than three months (fluctuations in the severity of the pain during this period are allowed)
* Ability to read and understand the English or Dutch language.

Exclusion Criteria:

* Surgery or invasive procedures within the last 3 months that can impact the physical activity level.
* Comorbidities: paresis and sensory disturbances with a neurological cause in the lower extremities, diabetes mellitus, autoimmune disorders, and all other non-musculoskeletal disorders that can produce pain and affect the physical activity level or physical functioning.
* Pregnancy or trying to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with one of the following musculoskeletal disorders: chronic low back pain (LBP); chronic neck pain (NP); chronic shoulder pain (CSP); osteoarthritis (OA); chronic Temporomandibular Disorder (CTMD); fibromyalgia (FM).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Global Physical Activity Questionnaire (GPAQ) | at baseline (cross-sectional)
  GPAQ collects information on physical activity participation in three settings (or domains) as well as sedentary behaviour and comprises of 16 questions (P1-P16). It allows categorization of the physical activity level of participants in either low, moderate, or vigorous. The domains are: Activity at work, Travel to and from places, and Recreational activities.
5 multiple choice questions based on The International Fitness Scale (IFIS) | at baseline (cross-sectional)
  This questioning evaluates 1) the perceived level of fitness of each participant in five subconstructs namely general physical fitness, cardiorespiratory fitness, muscular strength, speed/agility, and flexibility and 2) the perceived overall fitness level based on perceived physical ability in fictional daily situations.

SECONDARY OUTCOMES:
VAS-scores extracted from The Brief Pain Inventory short form (BPI-sf)(Q3-6) | at baseline (cross-sectional)
  This questionnaire evaluates the severity of a patient's pain and the impact of this pain on the patient's daily functioning. In Q3-6, the patient is asked to rate the worst, lowest, mean, and current pain intensity on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic pain.
Barriers to health quiz | at baseline (cross-sectional)
  The Barriers to Being Physically Active Quiz (18) is a 21-item measure assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely".
Physical Activity and Leisure Motivation Scale (PALMS) | at baseline (cross-sectional)
  the 40-item Physical Activity and Leisure Motivation Scale (PALMS) is designed to measure adult PA motivation. PALMS measures eight motives for participation in PA, namely mastery, enjoyment, psychological condition, physical condition, appearance, others' expectations, affiliation, competition/ego, on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The range of each PALMS sub-scale is 5 to 25 because each sub-scale has five items. The PALMS has been validated in previous studies.
Depression Anxiety Stress Scale (DASS-21) | at baseline (cross-sectional)
  This scale was developed to examine depression, anxiety and stress without the major impact of possible somatic factors. The questions can be answered with 0 (not at all or never applicable), 1 (a little or sometimes applicable), 2 (quite or often applicable) or 3 (very definitely or mostly applicable). A qualification score of 1-5 (normal to very severe) is calculated for each scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Fear-Avoidance Components Scale (FACS) | at baseline (cross-sectional)
  This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100).
Self-efficacy For Exercise (SEE) Scale | at baseline (cross-sectional)
  The Self-Efficacy for Exercise (SEE) scale is a revision of McAuley's self-efficacy barriers to exercise measure, a 13-item instrument that focuses on self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. This measure was developed initially for sedentary adults in the community who participated in an outpatient exercise program including biking, rowing, and walking. Prior research demonstrated sufficient evidence for reliability (alpha coefficient = 0.93) and validity, with efficacy expectations significantly correlated with actual participation in an exercise program.
PAREMO-20 | at baseline (cross-sectional)
  PAREMO-20 is a multidimensional instrument to determine the general rehabilitation-related motivation of the patients. PAREMO-20 consists of 20 items forming six subscales: "psychological burden", "physical burden", "social support","readiness to change", "knowledge", and "skepticism". Answers are given on a 4-point Likert scale. Higher values on subscales indicate higher rehabilitation motivation except for the subscale "skepticism". Here, higher scores indicate lower rehabilitation motivation.

OTHER OUTCOMES:
Modified Oswestry Disability Index (MODI) (only persons with chronic low back pain) | at baseline (cross-sectional)
  This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Neck Disability Index (NDI) (only persons with chronic neck pain) | at baseline (cross-sectional)
  The Neck Disability Index (NDI) is a questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic neck pain.
Shoulder Pain and Disability Index (SPADI) (only persons with chronic shoulder pain) | at baseline (cross-sectional)
  The SPADI is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with ADLs requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. This questionnaire is reliable and valid for use in persons with chronic low neck pain.
Fibromyalgia Impact Questionnaire (FIQR) (only persons with fibromyalgia) | at baseline (cross-sectional)
  The FIQR is a commonly used instrument in the evaluation of fibromyalgia (FM) patients. It has 21 individual questions. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'. the FIQR is divided into three linked sets of domains: (a) 'function' (contains 9 questions), (b) 'overall impact' (contains 2 questions), and (c) 'symptoms' (contains 10 questions).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) (only persons with osteorthritis) | at baseline (cross-sectional)
  The WOMAC is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), stiffness (2 items), and physical function (17 items).
TMD Disability Index (TDI) (only persons with chronic temporomandibular disorder) | at baseline (cross-sectional)
  The TMD Disability Index consists of ten questions regarding disability associated with CTMD, and each question is scored from 0-4. Higher scores represent greater levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, België, Belgium

IPD SHARING:
Plan to Share IPD: No